CLINICAL TRIAL: NCT00592891
Title: Oxygen Toxicity Effects Using Los-Pressure Hyperbaric Oxygen Therapy in the Treatment of Chronic Brain Injury
Brief Title: Oxygen Toxicity of HBOT in Chronic Brain Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paul G. Harch, M.D. (Other)
Collaborators: Harch Hyperbaric Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Paul G. Harch, M.D., Clinical Professor of Medicine, Louisiana State University Health Sciences Center in New Orleans
Organization: Louisiana State University Health Sciences Center in New Orleans (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSU IRB #5209
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Adult and Pediatric Chronic Cerebral Disorders
Keywords: brain injury; brain disorders
MeSH Terms: conditions — Brain Injuries; Brain Diseases | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperbaric oxygen therapy (Experimental): Patients undergoing low pressure HBOT for chronic brain injury
  Interventions: Drug: Hyperbaric oxygen therapy

INTERVENTIONS:
Drug: Hyperbaric oxygen therapy — Total body pressurized oxygen

SUMMARY:
Hypothesis: That HBOT can be toxic in the low-pressure range.

DETAILED DESCRIPTION:
The study is a retrospective review of the author's experience treating chronic brain injury with HBOT, supplemented by cases communicated to the author, who developed untoward effects during or after their HBOT. The object of the study was to affirm or refute the author's general impression that there was an optimal dose of HBOT in chronic brain injury which was lower than the traditional dose applied in chronic non-central nervous system wounding. Furthermore, when this lower dosage range was exceeded and approached the traditional doses for non-CNS wounding oxygen toxicity would result. To address these impressions the study seeks to review the author's medical records and other patient/doctor communications to the author where side effects of HBOT occurred in the treatment of chronic brain injury and abstract signs, symptoms, and the dose of HBOT employed.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral disorder of greater than one year's duration

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2002-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Oxygen toxicity | After completion of hyperbaric oxygen therapy

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Harch, M.D., Principal Investigator — LSU School of Medicine
Locations (1):
- Family Physicians Center, Marrero, Louisiana, United States